CLINICAL TRIAL: NCT06703034
Title: Characterization of the IFN-I Response in Subjects Who Experienced Severe or Mild Forms of COVID-19
Acronym: CARE-IF-COVID
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 69HCL24_0703; 2024-A01750-47 (Other: ANSM)
Record Dates: First submitted 2024-11-21; First posted 2024-11-25 (Actual); Last update posted 2025-06-15 (Actual); Status verified 2025-06

CONDITIONS: COVID-19
Keywords: COVID-19; interferon; disease severity; prognosis; Immune Functional Assays
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Intervention Model Description: This is a single-center, comparative, prospective, interventional study with minimal risk and constraints, RIPH category 2 outside of healthcare product
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mild patients (Other): Patients who experienced mild forms of COVID-19 during the first wave, without any prior vaccination, selected from the pre-existing COVID-Ser cohort (ClinicalTrial no. NCT04341142).
  Interventions: Other: Biological Sampling
- Severe patients (Other): Patients who experienced severe forms of COVID-19 during the first wave, without any prior vaccination, selected from the pre-existing NOSO-COR IMMUNO cohort (ClinicalTrial no. NCT04637867) and the RNIPH study (Research Not Involving Human Persons) named MIR-COVID.
  Interventions: Other: Biological Sampling

INTERVENTIONS:
Other: Biological Sampling — The procedures specifically carried out for the study during a single visit are as follows:
  * 1 nasopharyngeal swab for the baseline measurement of the nasal IFN-I score and to check for the presence of infection
  * Blood sample collection in:
  o1 yellow tube (5mL) for anti-interferon antibody measurement o1 PAXgene tube (2.5mL) for the baseline IFN score without stimulation o3 green heparin tubes (12mL) for performing immune-functional tests o2 large purple tubes (20mL) for biological collection (if the patient provides specific consent) oA total of 39.5mL of venous blood will be collected for the study during a single visit.
  * Stool collection at home by the patient, to be sent by mail to the Biological Resource Center (CRB) of the Hospices Civils de Lyon (HCL) within 10 days after the visit.
  * A food frequency questionnaire composed of 159 items measuring the frequency of consumption of foods and drinks over the past 12 months to complement the analysis of the gut microbiota.

SUMMARY:
Type I interferon (IFN-I) production is triggered by the detection of viral molecules, such as strands of viral RNA or DNA, by receptors known as PRRs (Pattern Recognition Receptors) present on many cell types. These interferons are secreted in minimal concentrations but can activate neighboring cells to secrete over 700 proteins with antiviral properties (inhibition of viral replication, destabilization of viral membranes, etc.). Thus, the IFN-I response serves as the immune system's first line of defense during a viral infection.

Very early in the COVID-19 pandemic, several research teams, including ours, identified a defect in the type I interferon response in about one in five subjects with severe COVID-19. In-depth studies have shown that 5 to 20% of these patients with severe COVID-19 disease have genetic mutations affecting genes involved in the activation cascade of the IFN-I pathway or produce autoantibodies that neutralize IFN-I, significantly impairing the effectiveness of their IFN-I response.

However, to date, not all causes of IFN-I response alteration are clearly identified, and 80% of patients suffering from severe COVID-19 do not appear to have evident genetic predispositions or anti-IFN-I autoantibodies, with the techniques currently available. This suggests the presence of other risk factors or causes that could potentially lead to alterations in the IFN-I response.

The gut microbiota is recognized for its influence on host health and immunity. SARS-CoV-2 (Severe Acute Respiratory Syndrome CoronaVirus 2) infection has been associated with altered gut microbiota and correlated with inflammatory and immune responses. However, the association between dysbiosis and IFN-I response has yet to be studied in humans.

Therefore, to improve the management of individuals affected by viral respiratory infections, it seems essential to explore alterations in the IFN-I response to identify individuals potentially at risk of developing severe forms. It is known that a failure in the IFN-I response in the early stages of a viral infection leads to uncontrolled viral replication, which may result in a severe form of the disease. Since this IFN-I response is essential for controlling all viral infections, regardless of the virus involved, the investigators hypothesize that this IFN-I deficiency could be responsible for severe infections from various respiratory viruses that may lead to severe forms, even though a direct association between IFN-I deficiency and higher mortality risk has only been reported for a few viruses, such as SARS-CoV-2 and influenza.

Furthermore, the investigators consider the possibility of other underlying causes of IFN-I deficiencies, distinct from the already observed anti-IFN-I autoantibodies and genetic mutations. To achieve this, the investigators hypothesize that the use of functional immune tests could reveal these other alterations.

By identifying these alterations in individuals, the investigators hope to more accurately predict their propensity to develop severe forms of viral infections.

Patients who experienced :

* mild forms of COVID-19 during the first wave, without any prior vaccination, selected from the pre-existing COVID-Ser cohort (ClinicalTrial no. NCT04341142)
* severe forms of COVID-19 during the first wave, without any prior vaccination, selected from the pre-existing NOSO-COR IMMUNO cohort (ClinicalTrial no. NCT04637867) and the RNIPH study (Research Not Involving Human Persons) named MIR-COVID (compliance with MR004 n°20_097_v2) could be recruited.

Biological samples will be collected specifically for the study, outside of a healthcare procedure. No biological sample in biocollections coming from COVID-ser and NOSO-COR IMMUNO studies and the RNIPH study (Research Not Involving Human Persons) named MIR-COVID will be used for this new protocol.

ELIGIBILITY:
Inclusion Criteria:

* Participant aged at least 18 years
* Previously included in the COVID-ser or NOSO-COR IMMUNO study as well as in the RNIPH study (Research Not Involving Human Persons) named MIR-COVID
* Weight of 50 kg or more

Exclusion Criteria:

* Current infection symptoms
* Immunosuppression defined by: bone marrow transplant within the past 24 months, chemotherapy within the past 6 months, HIV infection with CD4 <200/mm³ or <15%, corticosteroid therapy for more than 2 weeks with a daily dose over 10 mg of prednisolone equivalent, immunosuppressive treatment administered within the previous 3 months (6 months for rituximab), aplasia, asplenia, or splenectomy
* Pregnant, parturient, or breastfeeding woman
* Person deprived of liberty by judicial or administrative decision
* Person receiving psychiatric care
* Person admitted to a health or social institution for purposes other than research
* Person under guardianship or curators
* Person not affiliated with a social security scheme or similar coverage
* Patient participating in another ongoing interventional research study at inclusion"

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-12-02 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
IFN-I score measured post-stimulation by Influenza A virus (IAV) in vitro | At inclusion visit (Day 0)
  Comparison of the score IFN-I, measured by assessing the expression of a selection of IFN-I-stimulated genes, between the two groups of interest (mild or severe form).
  Given the limited advancement of studies on the interferon score following stimulation, no scoring scale is currently established. However, an increase in the score would be associated with a functional response to stimulation, indicating the absence of alterations in the targeted interferon induction pathway.

SECONDARY OUTCOMES:
IFN-I response induced post-stimulation in vitro by Poly I | At inclusion visit (Day 0)
  Comparison of the score IFN-I, measured by assessing the expression of a selection of IFN-I-stimulated genes, between the two groups of interest (mild or severe form).
  Given the limited advancement of studies on the interferon score following stimulation, no scoring scale is currently established. However, an increase in the score would be associated with a functional response to stimulation, indicating the absence of alterations in the targeted interferon induction pathway.
Induction of immune pathways post-stimulation at a transcriptomic/proteomic level on a panel of genes and cytokines/chemokines specifically involved in key processes of the immune response | At inclusion visit (Day 0)
  Comparison of gene expression levels, fold-changes expression, activation levels (Z-scores, p-value, FDR), and comparison of the concentrations of secreted cytokines/chemokines between the 2 groups of interest (mild or severe form)
Presence of anti-IFN-I autoantibodies | At inclusion visit (Day 0)
  Comparison of the presence and levels of anti-IFN-I autoantibodies between the two groups
Presence of other serum anti-cytokine autoantibodies detected by multiplex ELISA (Infinity Biomarker) | At inclusion visit (Day 0)
  Comparison of the presence and levels of other serum anti-cytokine antibodies between the two groups (mild or severe form)
Presence of genetic mutations affecting antiviral immune pathways | At inclusion visit (Day 0)
  Comparison of the frequency of genetic mutations affecting genes involved in the IFN-I response detected by sequencing between the two groups (mild or severe form)
Comparison of the blood and nasal IFN score in vivo without stimulation to the blood IFN score post-stimulation in vitro by the live attenuated Influenza A virus (IAV). | At inclusion visit (Day 0)
  Comparison of the blood and nasal IFN score in vivo without stimulation and the blood IFN score post-stimulation in vitro by the live attenuated Influenza A virus (IAV), Poly I:C, resiquimod (R848), diABZI, and IFNα
Propensity of individuals with a low IFN score post-stimulation by IAV to develop severe viral infections in the two winters following inclusion | After 2 winters (at last month 18)
  Correlation of the IFN score post-stimulation by IAV with severe infectious episodes during the two winters following inclusion
Overall composition of the gut microbiota and possibly the metabolome, depending on the intensity of the functional immune response post-stimulation. | At inclusion visit (Day 0)
  Correlation between the composition of the gut microbiota and possibly the metabolome and the immune response post-stimulation
IFN-I response induced post-stimulation in vitro by resiquimod (R848) | At inclusion visit (Day 0)
  Comparison of the score IFN-I, measured by assessing the expression of a selection of IFN-I-stimulated genes, between the two groups of interest (mild or severe form)
IFN-I response induced post-stimulation in vitro by diABZI | At inclusion visit (Day 0)
  Comparison of the score IFN-I, measured by assessing the expression of a selection of IFN-I-stimulated genes, between the two groups of interest (mild or severe form)
IFN-I response induced post-stimulation in vitro by IFNα | At inclusion visit (Day 0)
  Comparison of the score IFN-I, measured by assessing the expression of a selection of IFN-I-stimulated genes, between the two groups of interest (mild or severe form)
Comparison of the blood and nasal IFN score in vivo without stimulation to the blood IFN score post-stimulation in vitro by Poly I:C | At inclusion visit (Day 0)
  Comparison of the blood and nasal IFN score in vivo without stimulation and the blood IFN score post-stimulation in vitro by the live attenuated Influenza A virus (IAV), Poly I:C, resiquimod (R848), diABZI, and IFNα
Comparison of the blood and nasal IFN score in vivo without stimulation to the blood IFN score post-stimulation in vitro by resiquimod (R848) | At inclusion visit (Day 0)
  Comparison of the blood and nasal IFN score in vivo without stimulation and the blood IFN score post-stimulation in vitro by the live attenuated Influenza A virus (IAV), Poly I:C, resiquimod (R848), diABZI, and IFNα
Comparison of the blood and nasal IFN score in vivo without stimulation to the blood IFN score post-stimulation in vitro by diABZI | At inclusion visit (Day 0)
  Comparison of the blood and nasal IFN score in vivo without stimulation and the blood IFN score post-stimulation in vitro by the live attenuated Influenza A virus (IAV), Poly I:C, resiquimod (R848), diABZI, and IFNα
Comparison of the blood and nasal IFN score in vivo without stimulation to the blood IFN score post-stimulation in vitro by IFNα | At inclusion visit (Day 0)
  Comparison of the blood and nasal IFN score in vivo without stimulation and the blood IFN score post-stimulation in vitro by the live attenuated Influenza A virus (IAV), Poly I:C, resiquimod (R848), diABZI, and IFNα

CONTACTS AND LOCATIONS:
Locations (1):
- Hospices Civils de Lyon - Hôpital de la Croix-Rousse, Lyon, France

IPD SHARING:
Plan to Share IPD: Undecided